CLINICAL TRIAL: NCT05726877
Title: Determination of Optimal Positive End-expiratory Pressure in Prone Position During General Anesthesia Using Electrical Impedance Tomography in Pediatric Patient Under 17 Years of Age
Brief Title: Optimal PEEP in Pediatric Patients Under 17 Years of Age.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2208-091-1351
Record Dates: First submitted 2023-01-06; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Ventilation Therapy; Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): All patients will be enrolled in the same arm.
  Interventions: Other: ventilation strategy

INTERVENTIONS:
Other: ventilation strategy — Titrating positive end-expiratory pressure

SUMMARY:
This study aimed to investigate the differences in positive end-expiratory pressure titration in the supine and prone positions by age in pediatric patients under 17 years of age who received general anesthesia and then evaluate the hemodynamic stability.

ELIGIBILITY:
Inclusion Criteria:

* patients who are scheduled to undergo general anesthesia in the prone position
* patients who are in age under 17 years

Exclusion Criteria:

* had cyanosis or chronic respiratory failure
* had respiratory distress syndrome or bronchopulmonary dysplasia
* had laryngotracheal diseases
* had pulmonary hypertension
* receiving oxygen therapy

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Optimal positive end-expiratory pressure (PEEP) | 10 minutes after intubation
  result of decremental PEEP trial
Optimal positive end-expiratory pressure (PEEP) | 60 minutes after prone positioning
  result of decremental PEEP trial

SECONDARY OUTCOMES:
Impedance tidal variation | 10 minutes after intubation
  respiratory parameters measured by Electrical Impedance Tomography (EIT) device
Impedance tidal variation | 60 minutes after prone positioning
  respiratory parameters measured by EIT device
regional respiratory system compliance | 60 minutes after prone positioning
  respiratory parameters measured by EIT device
regional respiratory system compliance | 10 minutes after intubation
  respiratory parameters measured by EIT device
overdistension or atelectasis | 10 minutes after intubation
  respiratory parameters measured by EIT device
overdistension or atelectasis | 60 minutes after prone positioning
  respiratory parameters measured by EIT device
end-expiratory lung volume | 10 minutes after intubation
  respiratory parameters measured by EIT device
end-expiratory lung volume | 60 minutes after prone positioning
  respiratory parameters measured by EIT device
end-expiratory lung impedance | 10 minutes after intubation
  respiratory parameters measured by EIT device
end-expiratory lung impedance | 60 minutes after prone positioning
  respiratory parameters measured by EIT device
regional ventilation delay | 10 minutes after intubation
  respiratory parameters measured by EIT device
regional ventilation delay | 60 minutes after prone positioning
  respiratory parameters measured by EIT device
center of ventilation | 10 minutes after intubation
  respiratory parameters measured by EIT device
center of ventilation | 60 minutes after prone positioning
  respiratory parameters measured by EIT device
vital signs | 10 minutes after intubation
  blood pressure (mmHg)
vital signs | 60 minutes after prone positioning
  blood pressure (mmHg)
vital signs | 10 minutes after intubation
  oxygen saturation (%)
vital signs | 60 minutes after prone positioning
  oxygen saturation (%)
vital signs | 10 minutes after intubation
  heart rate (BPM)
vital signs | 60 minutes after prone positioning
  heart rate (BPM)
arterial blood gas analysis, if patients has arterial catheter | 10 minutes after intubation & 60 minutes after prone positioning
  oxygen and cardon dioxide tension

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, MD.Ph.D., Study Chair — Professor
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No